CLINICAL TRIAL: NCT06280521
Title: Validation en Langue française du Girls Questionnaire for Autism Spectrum Condition (fGQ-ASC) Chez Des Femmes Adultes
Brief Title: Validation of the Girls Questionnaire for Autism Spectrum Condition in French Langage
Acronym: fGQ-ASC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC23.0331
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Women with autistic spectrum disorder (Other)
  Interventions: Other: fGQ-ASC
- Men with autistic spectrum disorder (Other)
  Interventions: Other: fGQ-ASC
- Women without autistic spectrum disorder (Other)
  Interventions: Other: fGQ-ASC
- Men without autistic spectrum disorder (Other)
  Interventions: Other: fGQ-ASC

INTERVENTIONS:
Other: fGQ-ASC — French version of the Girl Questionnaire for Autism Spectrum Conditions (fGQ-ASC)

SUMMARY:
Autism spectrum disorders (ASD) are currently diagnosed at a rate of approximately 3 males per 1 female, while evidence suggests the rate may be 1.8 males per 1.2 females. It has been shown that affected women receive an autism diagnosis on average 5 years later than men. This delay is associated with deleterious consequences on the educational, psychological and physical health levels in these women. Currently, there are a number of obstacles that delay or prevent women with ASD from accessing diagnosis and specialized support. These include, in particular, gendered assumptions about how ASD manifests depending on the gender of the person concerned, a tendency for clinicians to attribute female autistic traits to causes other than ASD, measures of standardized ASD assessments that may not be sensitive enough to identify ASD females, and finally a demonstrated greater tendency among ASD females to camouflage or mask autistic traits in order to blend in in social situations. It is in this context that the Girl Questionnaire for Autism Spectrum Conditions (GQ-ASC) was developped and validated to address these fundamental gaps in the early identification and measurement of female ASD symptoms.

The GQ-ASC is presented as a self-questionnaire with 29 items which assess clinical characteristics specific to the adult female presentation of ASD in the dimensions (five) of imagination and play, camouflage, sensoriality, social situations and interests. To date, several studies have relevantly used the GQ-ASC in populations of adult ASD women, but none in French.

The main objective of this online study is therefore to measure the predictive validity of the French version of the Girl Questionnaire for Autism Spectrum Conditions (fGQ-ASC) for the diagnosis of ASD in adult women over 18 years of age and speaking French kindergarten. Subjects included in this online study will complete the protocol using any computer, tablet, or cell phone. We will include 400 participants (100 females-ASD, 100 females-nonASD, 100 males-ASD, 100 males-nonASD). This study will validate for the first time a screening tool for the diagnosis of ASD in women of French mother tongue over 18 years of age (the Girls Questionnaire for Autism Spectrum Condition French version - fGQ-ASC). This tool will have particularly significant benefits since it will help reduce the diagnostic delay among adult women with ASD in France and accelerate their access to specialized support.

DETAILED DESCRIPTION:
CONTEXT AND JUSTIFICATION OF THE RESEARCH Autism spectrum disorders (ASD) are currently diagnosed at a rate of approximately 3 males per 1 female, while evidence suggests the rate may be 1.8 males per 1.2 females. It has been shown that affected women receive an autism diagnosis on average 5 years later than men. This delay is associated with deleterious educational, psychological and physical health consequences in these women (Rynkiewicz & Łucka 2018).

Currently, there are a number of obstacles that delay or prevent women with ASD from accessing diagnosis and specialized support. These include, in particular, gendered assumptions about how ASD manifests depending on the gender of the person concerned, a tendency for clinicians to attribute female autistic traits to causes other than ASD, measures of standardized ASD assessments that may not be sensitive enough to identify ASD females, and finally a demonstrated greater tendency among ASD females to camouflage or mask autistic traits in order to blend in in social situations.

It is in this context that Attwood and colleagues (2011) developed the Girl Questionnaire for Autism Spectrum Conditions (GQ-ASC) to address these fundamental gaps in the early identification and measurement of female ASD symptoms. . In order to specifically and reliably assess the presentation of ASD in affected women, the initial stages and item development of this questionnaire were constructed and generated from the authors' extensive clinical expertise (Attwood et al. 2011). as diagnosticians. The questionnaire was then validated in English in adult women with ASD through rigorous analyzes (Brown et al. 2020).

The GQ-ASC is presented as a self-questionnaire with 29 items to be rated on a 4-point Likert scale (1 = Completely disagree, 2 = Mostly disagree, 3 = Mostly agree, 4 = Completely agree. agree) which assess clinical characteristics specific to the adult female presentation of ASD in the dimensions (five) of imagination and play, camouflage, sensoriality, social situations and interests. The original English version of the GQ-ASC makes it possible to identify 80.0% of women with ASD based on a cut-off score. This self-questionnaire also presents robust psychometric properties, including significant correlations between the five dimensions measured and with other questionnaires assessing ASD (Brown et al., 2020).

To date, several studies have relevantly used the GQ-ASC in populations of adult ASD women, but none in French. We make the main hypothesis that the French version of this questionnaire (fGQ-ASC) presents good predictive validity for the diagnosis of ASD in adult women over 18 years old and of French mother tongue. We also formulate the following hypotheses: 1) the fGQ-ASC presents poor predictive validity for the diagnosis of ASD in adult men over 18 years of age and of French mother tongue, 2) the fGQ-ASC scores are significantly higher higher in these women than in non-ASD women, ASD men and non-ASD men, 3) the fGQ-ASC presents satisfactory psychometric characteristics in adult ASD women over 18 years old and native speakers French.

PRIMARY OBJECTIVE The main objective of this study is to measure the predictive validity of the French version of the Girl Questionnaire for Autism Spectrum Conditions (fGQ-ASC) for the diagnosis of ASD in adult women over 18 years old and of French mother tongue. The fGQ-ASC is freely accessible and made available by the original authors. The fGQ-ASC was developed in 4 stages by the scientific leaders of the present study: 1) English to French online translation of the GQ-ASC (deepl.com), 2) rereading and possible modifications by 4 autistic adults (2 men and 2 women) of French mother tongue, 3) online back translation from French to English (deepl.com validated translation tool), 4) control and validation of the back translated version by the authors of the original version of the GQ-ASC.

MAIN JUDGMENT CRITERION Statistical significance of the chi-square test measuring the association between the following two categorical variables: 1) percentage of subjects in the female-ASD group presenting a suspected diagnosis of ASD according to the fGQ-ASC (total score ≥ 57) and 2) percentage of female ASD subjects with a diagnosis of ASD made by a doctor (Gold Standard). The women-ASD group is based on a distinction by birth sex.

SUMMARY DESCRIPTION OF THE STUDY DESIGN Subjects included in this online study will complete the protocol using any computer, tablet, or cell phone. No other material will be used. First, the information and non-opposition sheet is presented to the subject. If the subject agrees to participate in the study, he then completes the retrospective information according to his group which will make it possible to verify the inclusion criteria and then the self-questionnaires. The total completion time is estimated at 1 hour. The subject is free to take breaks during the examination if he wishes and to stop carrying out the research at any time if he wishes. The subject may also object to the use of their data after completion of the study by describing their request by email to the investigator and providing them with their random number provided during their participation in the study.

METHODOLOGY OF QUESTIONNAIRES / INTERVIEWS All the questionnaires in this study were validated in French, with the exception of the fGQ-ASC validated in English.

STATISTICAL ANALYSIS The analyzes will be carried out using R software once all the data has been collected. Descriptive statistics will include percentages of categorical variables and means and standard deviations of continuous variables. The measurement of the primary and secondary endpoints will be carried out with specific packages of the R software (lavaan and umx). The statistical significance threshold is set at p-value < 0.05.

The analyzes will be carried out by Dr Clément Dondé (PhD Neurosciences) and Adeline Lacroix (PhD Neurosciences).

INFORMATION RELATING TO RESEARCH IMPLEMENTATION

* Type of place where the research must take place: The subject included in this online study will carry out the protocol online via any computer, tablet or mobile phone, by connecting to the internet platform that hosts the study (https ://echoautism.org/). The subject will access it alone without the presence of an investigator.
* Estimated duration of the research: 2 years
* Estimated duration of participation per person: 1 hour maximum
* The research also involves the collection of retrospective data: age, sex, gender, family situation, place of life, level of study of the participant and that of the parents and professional situation will be collected for all the subjects; the presence of a comorbidity (neurodevelopmental, psychiatric, language delay), the age at diagnosis, the profession of the two professionals who made the diagnosis of ASD, the results of standardized diagnostic tests ADOS (Autism Diagnosis Observation Schedule) and ADI (Autism Diagnosis Interview), the presence of a language delay, the presence of a neurodevelopmental diagnosis other than ASD and the presence of an associated psychiatric diagnosis will be collected for subjects with ASD. The collection of this information does not allow the subject to be identified and does not present any particular risk to the subject.

PARTICIPANTS INCLUDED IN THE RESEARCH Number of participants interviewed: 400 (100 women-ASD, 100 women-nonASD, 100 men-ASD, 100 men-nonASD). Satisfactory size according to the recommendations of good practice for validation of scales.

Inclusion criteria:

* All groups: 18 years or older, French mother tongue
* ASD groups: have a diagnosis of ASD without intellectual development disorder (intellectual disability) made by professionals trained in autism
* Non-ASD groups: absence of diagnosis of psychiatric, neurological or neurodevelopmental disorder (including ASD made by professionals trained in autism), absence of suspicion of autism Secondary exclusion criteria: participant's wish to abandon the study currently being carried out.

Does the research include people without any conditions? Yes Methods of recruiting interviewees: Recruitment will be carried out by announcements sent by email to French university mailing lists and to online communities bringing together people with ASD. This method is the most effective for quickly informing a large number of individuals corresponding to the study inclusion criteria.

Information and traceability arrangements for non-opposition: An information sheet to be validated will be presented to each subject at the start of the study. The source data of each subject, the statistical analyses, as well as the final report of the study will be kept in an encrypted hard drive belonging to the CHU Grenoble Alpes and only accessible by the principal investigator for 15 years from the last date. visit of the last respondent included. This study does not include a consent form itself where the patient's identity would be recorded. Finally, as soon as the data of all respondents is transferred to the encrypted hard drive, the data will be permanently deleted from the internet platform hosting the study. The information collected during participation in the study will be treated in a strictly pseudonymized and confidential manner.

EXPECTED BENEFITS This study will validate for the first time a screening tool for the diagnosis of ASD in women of French mother tongue over 18 years of age (the Girls Questionnaire for Autism Spectrum Condition French version - fGQ-ASC). This tool will have particularly significant benefits since it will help reduce the diagnostic delay among adult women with ASD in France and accelerate their access to specialized support.

ELIGIBILITY:
Inclusion criteria:

* All groups: 18 years or older, French mother tongue
* ASD groups: have a diagnosis of ASD without intellectual development disorder (intellectual disability) made by professionals trained in autism
* Non-ASD groups: absence of diagnosis of psychiatric, neurological or neurodevelopmental disorder (including ASD made by professionals trained in autism), absence of suspicion of autism Secondary exclusion criteria: participant's wish to abandon the study currently being carried out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 50/50
Enrollment: 400 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
VP fGQ-ASC | baseline
  The main objective of this study is to measure the predictive validity of the French version of the Girl Questionnaire for Autism Spectrum Conditions (fGQ-ASC) for the diagnosis of ASD in adult women over 18 years old and of French mother tongue.

IPD SHARING:
Plan to Share IPD: Undecided